CLINICAL TRIAL: NCT03543202
Title: Comparison of Postoperative Analgesia and Patient Satisfaction of Unilateral Transversus Abdominis Plane (TAP) Block and Trocar Site Infiltration Anesthesia in Laparoscopic Cholecystectomy
Brief Title: Unilateral TAP Block vs Trocar Insertion Sites Infiltration Anesthesia in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Arik, Specialist in Anesthesia, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EmineTAP
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Biliary Disease
Keywords: Unilateral transversus abdominal plane block; Local infiltration anesthesia; Cholecystectomy; Postoperative analgesia
MeSH Terms: conditions — Gallbladder Diseases | interventions — Anesthesia, Local; Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: prospective randomised
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and outcome assesors will be blinded for the analgesia method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus abdominis plane block (Experimental): will receive 20ml bupivacaine for Transversus abdominis plane block and intravenous patient controlled analgesia
  Interventions: Drug: Transversus abdominis plane block; Drug: Intravenous patient controlled analgesia
- Local infiltration anesthesia (Active Comparator): will receive 20ml bupivacaine for Local infiltration anesthesia and intravenous patient controlled analgesia
  Interventions: Drug: local infiltration anesthesia; Drug: Intravenous patient controlled analgesia
- Intravenous patient control analgesia (Sham Comparator): will not receive any regional anethetic intervention will receive intravenous patient controlled analgesia
  Interventions: Drug: Intravenous patient controlled analgesia

INTERVENTIONS:
Drug: Transversus abdominis plane block — will receive 20ml bupivacaine for Transversus abdominis plane block and intravenous patient controlled analgesia
  Arms: Transversus abdominis plane block
Drug: local infiltration anesthesia — will receive 20ml bupivacaine for local infiltration anesthesia and intravenous patient controlled analgesia
  Arms: Local infiltration anesthesia
Drug: Intravenous patient controlled analgesia — will not receive any regional anesthetic intervention will receive intravenous patient controlled analgesia

SUMMARY:
Laparoscopic cholecystectomy is a commonly performed operation in general surgery practice. Peripheral nerve block methods commonly used for analgesia after this operation are: transversus abdominis plane block (TAP) and trocar insertion sites local anesthetic infiltration anesthesia In this study, we aimed to compare these methods in terms of postoperative analgesia, nausea-vomiting and patient satisfaction

DETAILED DESCRIPTION:
Patients will be randomly allocated by a computer generated random numbers list into three groups. After general anesthesia induction and intubation patients will receive analgesia according to group allocation. In group TAP (Group T) the transversus abdominis plane block will be commenced with ultrasound guidance while the patients is in the supine position with a subcostal approach using 20 mL 0.25% bupivacaine and 21 G block needle. In group infiltration anesthesia (Group I) the trocar insertion sites will be infiltrated with 20 mL 0.25% bupivacaine: 7 mL for the 10 mm trocar insertion sites and 3 mL for the 5 mm trocar insertion sites. The control group (Group C) will not receive any local anesthetic. All patients will receive rescue analgesia with intravenous patient controlled analgesia with tramadol (20 mg bolus dose and 20 minutes lockout time)

Postoperative pain will be assessed during resting and coughing with a Numeric Pain Scale (NRS) and nausea and vomiting with a Postoperative Nausea Vomiting Score at the postoperative 1, 3, 6, 12. and 24 hours. The amount of tramadol consumed in the postoperative period will be recorded. Patient satisfaction will be assessed with the Likert scale at postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of biliary disease

Exclusion Criteria:

* Uncooperative patients
* Blood coagulation disorders
* Laparatomy
* Obesity: body mass index >35
* Renal failure
* Hepatic failure
* Emergency surgery
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | Postoperative day 1
  Pain will be assessed with a 11 point numeric rating scale (0-10 whereas 0:no pain; 1-3: mild pain; 4-6: moderate pain and 7-10: severe pain)

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | Postoperative 1st hour, 3rd hour, 6th hour, 12th hour and 24th hour
  PONV will be assessed with a 5 point PONV intensity scale (1-4 whereas 1:absence of PONV; 2: nausea present, vomiting absent; 3 nausea present, vomiting once; 4: nausea present vomiting twice or more
Patient satisfaction | Postoperative 24 th hour
  Satisfaction will be assessed with a 5 point Likert scale (0-4 whereas 0:definitely disagree; 1:slightly agree; 3: agree; 4: strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Emine Arik, Dr, Principal Investigator — Ministry f Health
Locations (1):
- Diskapi Yıldırım Beyazıt EAH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chin KJ, McDonnell JG, Carvalho B, Sharkey A, Pawa A, Gadsden J. Essentials of Our Current Understanding: Abdominal Wall Blocks. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):133-183. doi: 10.1097/AAP.0000000000000545. PMID 28085788
- [Result] Bava EP, Ramachandran R, Rewari V, Chandralekha, Bansal VK, Trikha A. Analgesic efficacy of ultrasound guided transversus abdominis plane block versus local anesthetic infiltration in adult patients undergoing single incision laparoscopic cholecystectomy: A randomized controlled trial. Anesth Essays Res. 2016 Sep-Dec;10(3):561-567. doi: 10.4103/0259-1162.186620. PMID 27746552
- [Result] Ortiz J, Suliburk JW, Wu K, Bailard NS, Mason C, Minard CG, Palvadi RR. Bilateral transversus abdominis plane block does not decrease postoperative pain after laparoscopic cholecystectomy when compared with local anesthetic infiltration of trocar insertion sites. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):188-92. doi: 10.1097/AAP.0b013e318244851b. PMID 22330261
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789